CLINICAL TRIAL: NCT06256757
Title: Safety and Validity of Extracorporeal Fenestration and in Situ Fenestration in Patients With Aortic Disease Involving the Left Subclavian Artery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K2024031
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Aortic Dissection Aneurysm
MeSH Terms: conditions — Aortic Dissection | interventions — Fenestration, Labyrinth

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A（extracorporeal fenestration） (Experimental): Based on the preoperative CTA reconstructions, the diameter of the aorta and branch vessels, lengths, angles to the arch, clock positions, and related relationships are measured, and a preoperative design for the fenestrations is developed. The outer sheath of the stent graft is then pushed back for several centimeters under sterile conditions, allowing the proximal portion of the stent graft to be released. The length of the released segment should be one to two centimeters distal from the location of fenestration. Using a sterile ruler, the location of the fenestration is determined in accordance with the preoperative plan. The 12 o'clock position is considered to be at the front of the trigger. The position of the stent graft relative to the trigger is also referred to as the 12 o'clock position. If the fenestration must avoid stent struts, then the fenestration is deemed to be at 12 o'clock, as is the position of the trigger relative to the stent graft.
  Interventions: Procedure: fenestration
- B（In situ fenestration） (Sham Comparator): From the left brachial artery (LBA), a 6F angle-adjustable sheath (Lifetech, Inc., Shenzhen, China) is introduced retrogradely until its tip reaches the aortic stent graft. The tip is then adjusted to be as perpendicular as possible to the larger curve of the aortic stent graft. Once the sheath gets to the ideal position, a flexible needle (21 gauge, Futhrough, Lifetech, Inc.) is employed to create the fenestration in the aortic stent graft. Following the puncture, a 0.018-inch guidewire (V-18 ControlWire; Boston Scientific, Natick, MA) is inserted through the needle aperture and into the ascending aorta.
  Interventions: Procedure: fenestration

INTERVENTIONS:
Procedure: fenestration — Thoracic EndoVascular Aortic Repair (TEVAR) with fenestrations

SUMMARY:
This trial aims to demonstrate the safety and validity of extracorporeal fenestration and in situ fenestration in patients with aortic disease involving the left subclavian artery.

ELIGIBILITY:
Inclusion Criteria:(All of the following criteria were met for enrolment):

1. Patients aged greater than 18 years old and less than 80 years old.
2. Patients diagnosed with thoracic aortic disease, including thoracic aortic dissection, thoracic aortic aneurysm, thoracic aortic ulcer and intramural hematoma.
3. Patients needed endovascular repair (TEVER).
4. Patients who needed complete coverage of the left subclavian artery (planned landing Zone was in Zone 2 of the aortic zone).
5. The proximal lesion involved the proximal aorta within 1.5cm of the posterior edge of the left subclavian artery (LSA) opening, but not the left common carotid artery (LCCA).
6. Suitable femoral artery, iliac artery and brachial artery access can be used for endovascular treatment.
7. The patients could understand the purpose of the study, volunteered to participate in the study, and informed consent was signed by the subjects themselves or their legal representatives.
8. Patients were willing to undergo follow-up evaluation as required by the study protocol.
9. The life expectancy of the patient is more than 12 months.

Exclusion Criteria:(If any of the following criteria is met):

1. The lesion involved the proximal aorta of the LCCA opening (Zone 0 and Zone 1).
2. The patient has a definite connective tissue disease (e.g., Marfan syndrome).
3. The subjects had a history of previous thoracic endovascular aortic repair (TEVAR).
4. Patients who have had or may have had severe allergic reactions to contrast media (anaphylactic shock, exfoliative dermatitis, etc.).
5. Patients with contraindications to antiplatelet and anticoagulant drugs.
6. The patient's compliance was poor and the follow-up could not be expected on time.
7. Patients with acute systemic infection.
8. Patients cannot tolerate general anesthesia.
9. Patients judged by the investigator to be ineligible for endovascular treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 1 month postoperative
  all-cause mortality

SECONDARY OUTCOMES:
incidence of endoleak | postoperative (1, 6，12 months)
  incidence of endoleak
incidence of secondary intervention | postoperative (1, 6，12 months)
  incidence of secondary intervention
incidence of major adverse events (MAE) | postoperative (1, 6，12 months)
  incidence of major adverse events (MAE)
immediate technical success rate | immediate postoperative
  immediate technical success rate
all-cause mortality | postoperative (6, 12 months)
  all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Yanbo Lou, Study Director — The Fourth Affiliated Hospital Zhejiang University School of Medicine

IPD SHARING:
Plan to Share IPD: No
Upon reasonable request, the corresponding author will provide access to the full protocol, participant level-data and statistical code

REFERENCES:
- [Derived] Jia X, Wu J, Ding C, Lou Y. Safety and validity of extracorporeal fenestration and in situ fenestration in patients with aortic disease involving the left subclavian artery: a prospective, single-center, randomized controlled study. Trials. 2025 Jan 30;26(1):33. doi: 10.1186/s13063-025-08746-5. PMID 39885531